CLINICAL TRIAL: NCT01491373
Title: A Feasibility Investigation of Recombinant Human Bone Morphogenetic Protein-2 and Absorbable Collagen Sponge With LT-CAGE® Device for Anterior Lumbar Interbody Fusion in Patients With Degenerative Disc Disease
Brief Title: Pilot Study of rhBMP-2/ACS/LT-CAGE® for Anterior Lumbar Interbody Fusion in Patients With Degenerative Disc Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic Spinal and Biologics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-9504
Record Dates: First submitted 2011-12-12; First posted 2011-12-14 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2011-12

CONDITIONS: Degeneration of Lumbar Intervertebral Disc
Keywords: Degenerative Disc Disease; Symptomatic Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- rhBMP-2/ACS (Experimental)
  Interventions: Device: rhBMP-2/ACS/LT-CAGE® Device
- Autograft (Active Comparator)
  Interventions: Device: Autograft/LT-CAGE® Device

INTERVENTIONS:
Device: rhBMP-2/ACS/LT-CAGE® Device — rhBMP-2/ACS inserted into Sofamor Danek's LT-CAGE® device.
  Other Names: Recombinant human bone morphogenetic protein-2
  Arms: rhBMP-2/ACS
Device: Autograft/LT-CAGE® Device — LT-CAGE® device filled with autogenous bone taken from the patient's iliac crest
  Other Names: Autogenous bone graft
  Arms: Autograft

SUMMARY:
This study is designed to evaluate the feasibility of recombinant human bone morphogenetic protein-2 and absorbable collagen sponge with the tapered interbody fusion device (LT-CAGE® ) for anterior lumbar interbody fusion in patients with degenerative disc disease.

ELIGIBILITY:
Inclusion Criteria:

1. Has degenerative disc disease as noted by back pain of discogenic origin with degeneration of the disc confirmed by radiographic studies.
2. Has no greater than Grade 1 spondylolisthesis utilizing Meyerding's Classification (Meyerding HW, 1932.)
3. Has single level symptomatic degenerative involvement from L2 to S1.
4. Is between the ages of 18 and 65, inclusive, at the time of surgery.
5. Is willing to comply with the study plan and sign the Patient Informed Consent Form.
6. Has not responded to conservative treatment for a period of 5 months.
7. If of child-bearing potential, subject is non-pregnant (documented by a negative Pregnancy test within 72 hours of surgery), non-nursing female who agrees to use adequate contraception for 16 weeks following surgery

Exclusion Criteria:

1. Has spinal condition other than symptomatic degenerative disc disease at the involved surgical level.
2. Had previous anterior surgical procedures at the involved spinal level.
3. Has a condition which requires postoperative medications that interfere with fusion such as steroids or nonsteroidal anti-inflammatory drugs. (This does not include low dose aspirin for prophylactic anticoagulation.)
4. Has osteopenia, osteoporosis, or osteomalacia to a degree that spinal instrumentation would be contraindicated.
5. Has circulatory problems, such as thrombophlebitis, lymphedema, or vascular deficiency at the implant site.
6. Has symptomatic cardiac disease.
7. Has presence of active malignancy or history of cancer in the past 5 years.
8. Has overt or active infection.
9. Is obese, i.e., weight greater than 40% over ideal for their age and height.
10. Has fever (temperature > 101°F oral).
11. Has local inflammatory signs indicative of infection.
12. Has a documented metal allergy or intolerance.
13. Is involved in a worker's compensation or unresolved spinal litigation case.
14. Is mentally incompetent (either documented or in the opinion of the investigator).
15. Has psychogenic magnification of pain (in the opinion of the investigator).
16. Is a prisoner.
17. Is pregnant.
18. Is an alcohol and/or substance abuser.
19. Requires bone growth stimulation in the lumbar spine.
20. Is a tobacco user at the time of surgery.
21. Patient has received drugs which may interfere with bone metabolism within two weeks prior to the planned date of spinal fusion surgery (e.g., steroids or methotrexate).
22. Patient has a history of autoimmune disease (systemic lupus erythematosus or dermatomyositis).
23. The subject has a history of exposure to injectable collagen implants.
24. Patient's history includes hypersensitivity to protein pharmaceuticals (monoclonal antibodies or gamma globulins) or collagen.
25. Patient has received treatment with an investigational therapy within 28 days prior to implantation surgery or such treatment is planned during the 16 weeks following rhBMP-2/ACS implantation.
26. Patient has received any previous exposure to BMP.
27. The patient requires allograft or bone substitute as part of treatment.
28. Patient has history of endocrine or metabolic disorder known to affect osteogenesis (e.g. Paget's disease, renal osteodystrophy, Ehlers-Danlos syndrome, or osteogenesis imperfecta).
29. Patient in the physician's opinion, would not be a good candidate for this surgical procedure.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 1997-01; Primary Completion 1999-09 (Actual); Study Completion 1999-09 (Actual)

PRIMARY OUTCOMES:
Fusion | 24 month

SECONDARY OUTCOMES:
Pain Assessment (Oswestry Disability Index, ODI) | 24 month
Neurological Status Assessment | 24 month
Health status assessment (SF-36) | 24 month